CLINICAL TRIAL: NCT03958149
Title: Comparison of Measurements of the Cervical Spine in Adults With and Without Immobilisation
Brief Title: Measurements of Angulation of the C-spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Wellington Hospital (Other Government); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18SM4805; 19/SC/0059 (Other: Health Research Authority, Research Ethics Committee)
Record Dates: First submitted 2019-03-14; First posted 2019-05-21 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Cervical Spine
Keywords: Cervical spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal collar (Other): Participants will undergo MRI scans in and out a spinal collar to assess whether the measurements of angulation of the C-spine change whilst wearing a spinal collar.
  Interventions: Device: spinal collar

INTERVENTIONS:
Device: spinal collar — cervical collar to immobilise the cervical spine

SUMMARY:
This is a prospective study aiming to assess the shape of the neck in adults. In addition the study will look at the shape of the neck in a spinal collar and the comfort while wearing a spinal collar.

DETAILED DESCRIPTION:
The investigators aim to compare baseline scans of the neck in those aged 18yrs and older to a second neck scan where the participant is wearing a spinal collar. Experts will analyse the scans for measurements of angulations. In addition the study will collect demographic data and results from a validated patient questionnaire assessing comfort wearing the spinal collar.

The hypothesis:

1. The shape of the neck is different when comparing the young and old populations
2. The spinal collar does not alter the shape of the spine
3. The spinal collars are uncomfortable in the elderly population

ELIGIBILITY:
Inclusion Criteria:

1. Persons aged 18yrs and over to those aged 30yrs
2. Persons aged 70yrs and over
3. Ability to give informed consent to participate in the study

Exclusion Criteria:

1. Persons under 18yrs of age and those aged 31yrs -69yrs
2. Persons who lack capacity to consent for entry into the study
3. Persons who are unable to complete the visual analogue score or questionnaire due to co-existent visual and hearing loss. Severe hearing impairment will be defined as unable to hear the researcher with hearing aids if required. Severe visual impairment will be defined as being unable to read the patient information sheet even with visual aids.
4. Persons unable to understand the information leaflet in English.
5. Those with current neck pain, known previous C-spine injury or known medical condition affecting the spine.
6. Persons who do not pass the safety questionnaire to undergo an MRI scan
7. Persons who are unable to tolerate an MRI scan due to claustrophobia
8. Persons who are unable to transfer to the scanner table independently
9. Persons unable to lie flat and still for 10 minutes
10. Persons who do not give consent to their General Practitioner being informed of scan results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-04-13 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fertleman, Principal Investigator — Imperial College Healthcare NHS Trust/ The Wellington Hospital, London
Locations (2):
- United Kingdom (2):
  - The Wellington Hospital, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Young Group Aged 18-30 Years; Older Group Aged 70 Years and Over: Participants will undergo MRI scans in and out a spinal collar to assess whether the measurements of angulation of the C-spine change whilst wearing a spinal collar.
  Spinal collar: cervical collar to immobilise the cervical spine
Period: Overall Study
Arm/Group | Young Group Aged 18-30 Years | Older Group Aged 70 Years and Over
Started | 20 | 18
Completed | 20 | 17
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Young Group Aged 18-30 Years: Participants aged 18-30 years will undergo MRI scans in and out a spinal collar to assess whether the measurements of angulation of the C-spine change whilst wearing a spinal collar.
  Spinal collar: cervical collar to immobilise the cervical spine
- Older Group Aged 70 Years and Over: Participants aged 70 years and older will undergo MRI scans in and out a spinal collar to assess whether the measurements of angulation of the C-spine change whilst wearing a spinal collar.
  Spinal collar: cervical collar to immobilise the cervical spine
- Total: Total of all reporting groups
Arm/Group | Young Group Aged 18-30 Years | Older Group Aged 70 Years and Over | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Full Range); unit: years] | 25.3 [21 to 30] | 77.3 [71 to 102] | 51.8 [21 to 102]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 18 | 38
Visual analogue scale of pain [Mean (Full Range); unit: units on a scale] — 'Visual Analogue Scale' for pain (self reported: minimum 0=no pain at all, maximum 10= worst pain imaginable)
  units on a scale | 0.75 [0.0 to 5.0] | 0.87 [0 to 5.1] | 0.81 [0 to 5.1]

OUTCOME MEASURES:

1. Primary Outcome: Measurements of Angulation of the Neck (C-spine) on MRI Scans
Description: Comparison of the measurements of angulation of the neck (assessed on MRI imaging) in the young person compared to the older person. Statistical analysis to allow comparison of groups.
Time Frame: Baseline MRI image, approximately 30 minutes and second MRI image (with collar on), after one hour of wearing collar.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Measurements of Angulation of the Young Group Neck (C-spine); Measurements of Angulation of the Older Group Neck (C-spine): Baseline angles: Total lordosis angle, Upper cervical lordosis angle, Lower cervical lordosis angle, T1 slope angle, Neck tilt angle, Thoracic inlet angle and the Individual vertebral angles from C1 to T2.
Arm/Group | Measurements of Angulation of the Young Group Neck (C-spine) | Measurements of Angulation of the Older Group Neck (C-spine)
Number analyzed (Participants) | 20 | 17
degrees
  Total lordosis angle | 10.6 (8.7) | 21.6 (11.9)
  Upper cervical lordosis angle | 5.5 (4.0) | 4.1 (3.5)
  Lower cervical lordosis angle | 9.9 (6.9) | 18.7 (11.7)
  T1 slope angle | 62.4 (5.6) | 54.6 (9.5)
  Neck tilt angle | 44.0 (10.3) | 52.8 (13.5)
  Thoracic inlet angle | 106.4 (10.9) | 107.4 (20.1)
  Individual vertebral angle of C1 | 0.5 (11.3) | 0.2 (6.2)
  Individual vertebral angle of C2 | 1.5 (7.0) | -1.0 (4.6)
  Individual vertebral angle of C3 | -1.3 (6.1) | -0.6 (3.5)
  Individual vertebral angle of C4 | -2.4 (7.1) | -1.4 (3.8)
  Individual vertebral angle of C5 | -2.2 (8.8) | -1.3 (4.0)
  Individual vertebral angle of C6 | -0.9 (9.7) | -4.5 (2.9)
  Individual vertebral angle of C7 | -1.3 (10.9) | -5.0 (6.2)
  Individual vertebral angle of T1 | -0.3 (9.5) | -5.6 (6.5)
  Individual vertebral angle of T2 | -0.9 (11.1) | -3.8 (7.0)
Statistical Analysis 1: Comparison: Measurements of Angulation of the Young Group Neck (C-spine) vs Measurements of Angulation of the Older Group Neck (C-spine); Test type: Superiority; p < 0.001, Independent t-test

2. Secondary Outcome: The Degree of Change in Measurements of Angulation of the Neck (C-spine) on MRI Scans Whilst Wearing a Spinal Collar Compared to When Not Wearing a Spinal Collar.
Description: Comparison of the degree of change of measurements of angulation of the neck from MRI scans of a young persons neck (C-spine) in and out of a spinal collar to those of an older persons neck (C-spine) in and out of a spinal collar on MRI imaging. Statistical analysis to allow comparison of groups.
Time Frame: Baseline MRI image, approximately 30 minutes and second MRI image (with collar on), after one hour of wearing collar.
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Change in Degree of Angulation of the Young Group Neck (C-spine); Change in Degree of Angulation of the Older Group Neck (C-spine): Change in degree of angle from pre-collar status to post-collar status: Individual vertebral angles from C1 to T2.
Arm/Group | Change in Degree of Angulation of the Young Group Neck (C-spine) | Change in Degree of Angulation of the Older Group Neck (C-spine)
Number analyzed (Participants) | 20 | 17
degrees
  Individual vertebral angles of C1 | 0.14 (0.16) | 0.12 (10.80)
  Individual vertebral angles of C2 | 0.11 (0.15) | 0.73 (9.24)
  Individual vertebral angles of C3 | 0.1 (0.2) | 4.8 (7.7)
  Individual vertebral angles of C4 | 0.2 (0.1) | 10.7 (6.1)
  Individual vertebral angles of C5 | 0.2 (0.1) | 14.7 (7.1)
  Individual vertebral angles of C6 | 0.2 (0.1) | 15.9 (6.9)
  Individual vertebral angles of C7 | 0.2 (0.1) | 18.7 (8.9)
  Individual vertebral angles of T1 | 0.2 (0.1) | 16.5 (9.4)
  Individual vertebral angles of T2 | 0.2 (0.1) | 16.1 (11.9)
Statistical Analysis 1: Comparison: Change in Degree of Angulation of the Young Group Neck (C-spine) vs Change in Degree of Angulation of the Older Group Neck (C-spine); Test type: Superiority; p < 0.05, Factorial Mixed ANOVA

3. Other Pre Specified Outcome: Level of Comfort in and Out of a Spinal Collar.
Description: Comfort after one hour of wearing a spinal collar measured by the 'Visual Analogue Scale' for pain (self reported: minimum 0=no pain at all, maximum 10= worst pain imaginable)
Time Frame: Baseline, approximately 30 minutes and after wearing a collar for one hour
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Older Group Aged 70 Years and Over: Participants aged 70 years and over will undergo MRI scans in and out a spinal collar to assess whether the measurements of angulation of the C-spine change whilst wearing a spinal collar.
  Spinal collar: cervical collar to immobilise the cervical spine
Arm/Group | Young Group Aged 18-30 Years | Older Group Aged 70 Years and Over
Number analyzed (Participants) | 20 | 17
units on a scale | 2.91 [0 to 8.7] | 1.35 [0 to 5.7]

ADVERSE EVENTS:
Time Frame: Duration of time whilst actively participating in study (1 day)
Arm/Group | Young Group Aged 18-30 Years | Older Group Aged 70 Years and Over
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT03958149/Prot_SAP_000.pdf